CLINICAL TRIAL: NCT07156591
Title: Impact of Neuropathy on the Risk of Semaglutide-Induced Gastric Retention: A Single-Center, Prospective, Observational Study
Brief Title: Impact of Neuropathy on the Risk of Semaglutide-Induced Gastric Retention
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: 2025K249
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Gastric Retention
Keywords: Semaglutide; Gastric Retention; Esophagogastroduodenoscopy; Diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Diabetic patients with neuropathy receiving uninterrupted semaglutide therapy
  Interventions: Procedure: Esophagogastroduodenoscopy
- Non-exposure group: Diabetic patients without neuropathy receiving uninterrupted semaglutide therapy
  Interventions: Procedure: Esophagogastroduodenoscopy

INTERVENTIONS:
Procedure: Esophagogastroduodenoscopy — Assess the gastric retention during esophagogastroduodenoscopy

SUMMARY:
A prospective, single-center, observational study to compare the risk of gastric retention between the exposure group (with neuropathy) and non-exposure group (without neuropathy) in diabetic patients receiving uninterrupted semaglutide therapy

DETAILED DESCRIPTION:
Glucagon-like peptide-1 receptor agonists (GLP-1RAs) exert their effects by mimicking the action of endogenous GLP-1, activating GLP-1 receptors located in the pancreas, brain, and gastrointestinal tract. On one hand, they promote insulin secretion and suppress glucagon release; on the other, they reduce gastrointestinal motility and delay gastric emptying by stimulating the sympathetic nervous system and inhibiting the parasympathetic nervous system, including enhancing pyloric sphincter contraction. Through these dual mechanisms, GLP-1RAs improve glycemic control and facilitate weight management in patients with type 2 diabetes mellitus (T2DM).

Multiple prior studies and recent meta-analyses have shown that continuous use of GLP-1RAs increases the risk of gastric retention, potentially leading to aspiration and significantly elevating anesthesia-related risk. As a result, several recent expert consensus statements and clinical guidelines-including the 2023 ASA Expert Consensus and the 2025 ASGE Clinical Guidelines-recommend that weekly GLP-1RAs be discontinued for at least one week prior to procedures requiring anesthesia, regardless of dosage. For patients whose discontinuation interval is less than one week, preoperative gastric ultrasound is advised to rule out gastric retention; otherwise, anesthesia should proceed under a "full stomach" protocol.

Given the close connection between GLP-1RA pharmacodynamics and both the autonomic and peripheral nervous systems-and considering that neuropathy is one of the most prevalent complications in T2DM patients-a previous study explored the role of diabetic neuropathy in GLP-1RA-induced delayed gastric emptying. Interestingly, it found that GLP-1RA use in diabetic patients with neuropathy did not significantly slow gastric emptying. However, this study was limited by a small sample size and did not evaluate the actual risk of gastric retention, limiting its clinical relevance.

To further investigate the impact of neuropathy on GLP-1RA-induced gastric retention, we propose a single-center, prospective, observational study. Semaglutide, the most widely used weekly GLP-1RA, will be selected as the study drug. The study will enroll T2DM patients with or without diabetic neuropathy who have been on long-term semaglutide therapy (≥4 weeks) prior to undergoing upper endoscopy. The primary objective is to assess the risk of gastric retention under endoscopic examination.

The findings of this study may contribute to more personalized perioperative management strategies for diabetic patients on semaglutide, potentially reducing anesthesia-related risks while minimizing the glycemic instability associated with prolonged drug discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of diabetes mellitus.
* Long-term use of semaglutide (for at least 4 weeks) without discontinuation prior to endoscopic examination.
* Age ≥ 18 years, with no restriction on sex.
* American Society of Anesthesiologists (ASA) physical status classification I-II.
* Fasting for at least 8 hours and no water intake for at least 4 hours prior to gastroscopy.
* Underwent assessment for both autonomic and peripheral neuropathy within 2 weeks prior to gastroscopy, with a clear determination of neuropathy status.

Exclusion Criteria:

* History of hiatal hernia or any prior gastric surgery (including gastrectomy, Roux-en-Y gastric bypass, etc.).
* Pregnancy.
* Medically unfit for gastrointestinal endoscopy.
* Deemed unsuitable for participation at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients undergoing esophagogastroduodenoscopy who have been on long-term semaglutide therapy (≥4 weeks), either with neuropathy (exposure group) or without neuropathy (non-exposure group).
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Rate of gastric retention | immediately after the esophagogastroduodenoscopy
  Gastric retention was defined as the presence of solid residues in the stomach or liquid retention exceeding 1.5 mL/kg

SECONDARY OUTCOMES:
Gastric Mucosal Visibility Score | immediately after the esophagogastroduodenoscopy
Rate of hypoxemia and aspiration events | immediately after the esophagogastroduodenoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital, Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)